CLINICAL TRIAL: NCT00309114
Title: Prevention of UTI in Persons With Spinal Cord Injury
Brief Title: Prevention of Urinary Tract Infection (UTI) in Persons With Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rabih Darouiche, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5R01HD043943-03 (NIH); H-8393 (Other: Baylor College of Medicine)
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infections
Keywords: UTI; SCI; E coli; Prevention
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections | interventions — Antibiosis

STUDY DESIGN:
Intervention Model Description: Active intervention that includes bacterial interference using E. coli 83972 is compared with a placebo intervention.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventions for Experimental Arm (Experimental): Bacterial Interference with Escherichia coli 83972. Each bladder inoculation contains the study organism, E. coli 83972, suspended as a clear solution in sterile physiological saline.
  Interventions: Procedure: bacterial interference
- Interventions for Control Arm (Placebo Comparator): Each bladder inoculation contains sterile physiological saline that does not contain the study organism.
  Interventions: Procedure: bacterial interference

INTERVENTIONS:
Procedure: bacterial interference

SUMMARY:
Urinary tract infection (UTI) is the most common infection in patients with spinal cord injury (SCI) and is linked to major undesired results or complications including death. The bladder of SCI patients, especially those with indwelling catheters, is usually colonized by bacteria, some of which do and others which do not cause symptoms of UTI. Bacteria that do not cause symptoms are often called benign colonizers and are often left untreated because they may provide some protection against infection with more harmful bacteria. This idea of using benign bacteria to prevent infections with symptoms is called bacterial interference. A prototype strain, Escherichia coli 83972, was shown to begin and continue for extended periods of time non symptom causing colonization of the human bladder and to hold back symptom causing infections of the neurogenic bladder. Data from pilot studies at two medical centers indicated that bacterial interference might be a useful therapy for reducing the rate or frequency of UTI in SCI patients. Because almost all SCI patients have a UTI at some time, and also the large costs of treating this infection, studying the impact of bladder colonization with E. coli 83972 on the rate of symptom causing UTI has an amazing potential for improving the quality of life of SCI patients and decreasing the cost of health care. Like with other preventive plans such as vaccination, for instance, it is important to explore the effectiveness of this new preventive approach. The project is a prospective, randomized, double blind, multi-center study that deals with specific pieces of bacterial interference in SCI patients.

HYPOTHESES: Placing non symptom causing bacteria (E. coli 83972) into SCI patients' bladders reduces the rate of symptom causing UTI.

A. SPECIFIC AIM: Determine how bladder colonization with E. coli 83972 or similar bacteria affects the rate of symptom causing urinary tract infections in a large group of SCI and Spina Bifida patients by conducting a prospective, randomized, placebo-controlled, multi-center clinical trial.

DETAILED DESCRIPTION:
This clinical trial will be take place in a total of 7 medical centers that care for Spinal cord injury (SCI) and Spina Bifida patients. A total of 160 patients will be allowed to take part in the study.

The study coordinator will interview patients by telephone and in person who express an interest in taking part in the study. After an informed consent and HIPAA documents are reviewed and all of the patients questions are answered, then they will be asked to sign these two forms. Then a code number will be assigned to each patient and used along with their initials to identify them for the remainder of the study. All study participants will have a complete history and physical examination including ASIA classification, serum creatinine and a urine culture immediately upon entry into the study. One of the following 3 diagnostic tests must be completed within the 3 months before the study: KUB, IVP, or non-contrast abdominal CT scan. A voiding cystourethrogram with fluoroscopy (VCUG) alone or as part of a video urodynamics evaluation must be completed within 1 year before the study.

Randomization and sample size: Enrolled subjects will be randomized in a 3:1 ratio to receive bladder inoculation either with E. coli 83972 (experimental group) or with placebo (control group). This randomization ratio was selected because around 1/3 of colonized subjects are expected to remain colonized for 12 months.

Bladder inoculation: At study entry, a urine culture and sensitivity test will be completed using a fresh mid stream (after the urine is flowing) urine sample removed via a catheter into the bladder. Subjects will stop all actions to prevent or slow urinary tract infection (UTI) for at least two weeks upon entry into the study. Each subject will be treated with correct antibiotics for 7 - 10 days and any existing urinary catheter changed three days after starting antibiotic treatment. Forty-eight to 72 hours or (80 to 90 hours for fluoroquinolone antibiotics) after completion of antibiotics, the urine will be re-cultured and the lower urinary tract inoculated with E. coli 83972 or placebo.

Most subjects, even those with external condom catheters, have worn a Foley catheter at some time, and would be expected to know the catheter size that best fits them. Subjects will be inoculated on three consecutive days. Inoculation will consist of putting into the bladder via a sterile catheter 10 ml of normal saline alone or containing E. coli 83972. Subjects who are incontinent at low bladder volumes will be monitored with a Foley catheter balloon blocking the bladder neck or diversion stoma for 30 minutes after inoculation. After 30 min., the clamp will be released and the bladder allowed to drain for an additional 30 min. The bladder inoculation will be repeated a second time unless an unexpected adverse event (complication) is encountered. After the catheter is un-clamped for the second time, the subject will be observed for 30 min. before discharge.

If the 48-hour culture from the sample taken just prior to inoculation is positive for bacteria, and E. coli 83972 colonization was not present in the sample, another antibiotic treatment/inoculation cycle will be attempted. The timing of the second attempt will be decided by the CORE director and the local principal investigator. At the correct time, another 7-10 day course of antibiotic therapy will be repeated. Three days after starting antibiotics, any existing urinary catheter will be changed. Forty-eight to 72 hours or (80 to 90 hours for fluoroquinolone antibiotics) after completion of this course of antibiotics, the urine will be re-cultured and then the bladder re-inoculated. If the 48 hour culture taken just prior to this inoculation is again positive for any bacteria other than E. coli 83972, and E. coli 83972 colonization is not present as a result of the second inoculation cycle, a third cycle of antibiotic treatment/inoculation will be attempted. The timing of the 3rd attempt will be decided by the CORE director and the local principal investigator. No further colonization attempts will be made in study participants who are not colonized after three sets of attempts. We will continue to monitor subjects in this group for the remaining months of the study, but for analysis purposes, they will be treated as "never colonized".

All inoculated subjects who remain without symptoms will return to their study center to have a urine sample collected and a brief medical interview one week after inoculation and monthly for the remaining 12 months. The CORE director can allow a subject who lives far from any center to mail their monthly urine samples directly to the CORE. All needed supplies such as: urine specimen containers, proper shipping containers, labels, pre-paid postage, etc.… will be provided at no cost to the subject. The subject's study site will contact them to conduct the brief medical interview.

At the end of 12 months, subjects will receive an antibiotic to clear E. coli 83972 from their bladder and the study will be finished. If a subject experienced an adverse event (something unexpected) during the study, they will be followed by the research staff until the event has gone back to normal or resolved.

Growth of E. coli 83972 in the urine will indicate bladder colonization. Subjects will be considered colonized as long as E. coli 83972 is present and even if there are other bacteria in the urine. Subjects who develop symptoms of a UTI will be treated with proper antibiotics guided by susceptibility patterns for the bacteria(s) grown from urine cultures. Urine cultures collected prior to starting treatment will be tested for E. coli 83972. It is important to note that although the method of bladder inoculation carries some risk of causing symptoms of a UTI, that risk is rather small and will be shared by all subjects.

There exists a risk that clamping of the bladder for 30 minutes may result in autonomic dysreflexia in some patients, especially those who dump urine. All subjects will be asked about a history of autonomic dysreflexia or any unexpected response to bladder filling prior to inoculation. Before beginning inoculation, urodynamics data will be reviewed. All subjects with a lesion level above T7 will have their blood pressure (BP) monitored every 3 - 5 minutes while the catheter is clamped. If the subject reports any symptoms associated with autonomic dysreflexia; e.g., headache, sweating, flushing and so forth, or if the BP monitor records a systolic or diastolic BP 20 mm Hg above baseline or in any case, if the systolic BP exceeds 150 or the diastolic BP exceeds 100 mm Hg, the catheter will be un-clamped. Monitoring will continue until the subject is without symptoms with their baseline BP's. Interventions, including elevating the head of the bed, lowering the legs, as well as pharmacologic measures (nitropaste, nifedipine, etc.) will be used if needed. The use of pharmacologic measures and any other measures will follow the Clinical Procedures Guidelines for acute management of autonomic dysreflexia published by the Paralyzed Veterans of America.

ELIGIBILITY:
Inclusion Criteria:

* 15 years or older
* Living in institutional or non-institutional settings
* 6 months post spinal cord injury (SCI) prior to entry or have Spina Bifida
* Loss of bladder function
* Loss of normal bladder sensation
* Selected in-patients involved in the Rehab I program
* Catheter dependent, having either an indwelling urinary catheter or using an external catheter, intermittent catheterization, or vesical urinary diversion (original bladder, whole or in part, serves as the collection receptacle for urine) for bladder management.
* Two or more urinary tract infections (UTI) within the 12 months prior to the study.
* Capable of understanding the purpose of the study and providing informed consent to participate
* Pursue appropriate follow-up over the course of the study.

Exclusion Criteria:

* Any bladder stone(s)
* Kidney stone(s) greater than 1 cm in size
* Any obstructing kidney stone regardless of size
* Nephrostomy tube(s)
* Supravesical diversion (original bladder is no longer part of the collection receptacle for urine)
* Congenital genitourinary anomaly that predisposes to UTI
* Conditions anticipated to require recurrent antibiotic therapy for extraurogenital infection (e.g., recurrent pneumonia, decubitus ulcer)
* Current immunosuppression
* Vascular prosthesis
* Congenital or acquired cardiac disease susceptible to vegetative infections
* Bladder capacity of less than 50 cc
* Individuals with known significant cognitive impairment resulting from trauma, disease, or congenital conditions
* Women of childbearing age who engage in unprotected intercourse
* Women who are currently pregnant will be included in the study
* Women who become pregnant during the study will be discontinued from participation. Pregnant women who experience UTI or prolonged asymptomatic bacteriuria are at risk of bearing infants with low birth weight.
* Children
* Prisoners
* Men and women with significant known mental illness or emotional disorders related to organic or inorganic causes.

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2004-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Putting E. coli 83972 into the bladder of SCI patients reduces the rate of symptomatic UTI. | 12 Months

SECONDARY OUTCOMES:
Study the affect of bladder colonization with E. coli 83972 on the rate of symptom causing UTI in a large group of SCI and Spina Bifida patients. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Darouiche, MD, Principal Investigator — Baylor College of Medicine; Barbara Trautner, MD, PhD, Study Director — Baylor College of Medicine
Locations (5):
- United States (5):
  - Shepherd Center, Atlanta, Georgia
  - Rehab Institute Chicago, Chicago, Illinois
  - UT Southwestern, Dallas, Texas
  - Michael E Debakey VA Medical Center, Houston, Texas
  - The Institute for Rehabilitation and Research (TIRR), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darouiche RO, Thornby JI, Cerra-Stewart C, Donovan WH, Hull RA. Bacterial interference for prevention of urinary tract infection: a prospective, randomized, placebo-controlled, double-blind pilot trial. Clin Infect Dis. 2005 Nov 15;41(10):1531-4. doi: 10.1086/497272. Epub 2005 Oct 13. PMID 16231269
- [Background] Darouiche RO, Donovan WH, Del Terzo M, Thornby JI, Rudy DC, Hull RA. Pilot trial of bacterial interference for preventing urinary tract infection. Urology. 2001 Sep;58(3):339-44. doi: 10.1016/s0090-4295(01)01271-7. PMID 11549475
- [Background] Hull R, Rudy D, Donovan W, Svanborg C, Wieser I, Stewart C, Darouiche R. Urinary tract infection prophylaxis using Escherichia coli 83972 in spinal cord injured patients. J Urol. 2000 Mar;163(3):872-7. PMID 10687996
- [Result] Darouiche RO, Green BG, Donovan WH, Chen D, Schwartz M, Merritt J, Mendez M, Hull RA. Multicenter randomized controlled trial of bacterial interference for prevention of urinary tract infection in patients with neurogenic bladder. Urology. 2011 Aug;78(2):341-6. doi: 10.1016/j.urology.2011.03.062. Epub 2011 Jun 17. PMID 21683991